CLINICAL TRIAL: NCT03846037
Title: Effects of Proprioceptive Exercises Associated With Vibratory Stimuli on Electromyographic Activity, Postural Oscillation and Sense of Joint Position in Healthy Individuals
Brief Title: Evaluation of the Balance, Muscular Electric Activity, Proprioception Before and After in the Vibratory Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 18643413.3.0000.5503
Record Dates: First submitted 2019-02-11; First posted 2019-02-19 (Actual); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Therapeutics
Keywords: Proprioception; Balance; Whole-body Vibation; One-foot Stance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ground (Placebo Comparator): Participants in this group perform protocol exercises on a stable surface.
  Interventions: Other: Proprioceptive exercise on the ground (stable surface)
- vibrating platform (Experimental): Participants in this group perform protocol exercises on a vibrating platform.
  Interventions: Other: Proprioceptive exercise on the vibratory platform

INTERVENTIONS:
Other: Proprioceptive exercise on the vibratory platform — Unipodal support over the non-dominant lower limb with the contralateral limb in a knee flexion near 90ºon the vibratory platform
  Arms: vibrating platform
Other: Proprioceptive exercise on the ground (stable surface) — Unipodal support over the non-dominant lower limb with the contralateral limb in a knee flexion near 90ºon the ground
  Arms: Ground

SUMMARY:
Introduction: Proprioception refers to the information's dynamic, sent to central nervous system by the free nerve endings and mechanoreceptors, about the biomechanics relationship for the joint tissue. The proprioceptive exercises show a big prophylactic action by musculoskeletal injuries. Among the top modalities of these exercises, it can be cited the Whole Body Vibration (WBV). Objectives: The objective of this study was to evaluate and compare the joint position sense, muscle electric activity and the postural sway in healthy individuals, before and after performing proprioceptive exercises on the vibrational platform or on a stable surface. Materials and Methods: 20 healthy young (24,85 + 4,27 years) were recruited, randomly divided into two groups, Control Group (GC) and Experimental Group (GE). Were realized evaluates of the proprioception by means of the joint position sense, the muscle electric activity of peroneus longus, gastrocnemius medialis, vastus medialis and gluteus medium, and the postural sway by means of the postural sway before and after one assistance consisting of 4 sets of 60s with unipodal standing position on soil (GC) or on vibrational platform (GE).

DETAILED DESCRIPTION:
The individuals who composed the two groups performed the same exercise protocol, however, on different surfaces:

* Control group: stable surface.
* Experimental group - vibratory platform, make / model Nissan Fisio; orbital amplitude: 6 mm; frequency: 30 Hz The exercises consisted of unipodal support on the non-dominant lower limb with the contralateral limb in a knee flexion near 90º. This exercise is a proprioceptive test that requires more than all joints and musculature of the lower limb, and is widely used in studies, for providing obvious clinical signs in the presence of dysfunctions.

Activities were performed with the individual standing without using any type of footwear, remaining without support of the hands and with the upper limbs abducted to 90º with the fixed eye on the horizon line. Both groups performed 4 sets of 60s of sustained posture. In the intervals between the series there was the rest of 60s, remaining in orthostasis with support of the upper limbs.

ELIGIBILITY:
Inclusion Criteria:

* Individuals from 18 to 30 years;
* Healthy;
* Sedentary;
* That they agree with the Free and Informed Consent Term.

Exclusion Criteria:

* Recent surgery;
* Open wounds;
* Contagious skin diseases;
* Glaucoma;
* Labyrinthitis;
* Uncontrolled heart diseases;
* Pacemaker;
* Lower limb injuries;
* Neurological dysfunctions;
* Pain in the lower limbs;
* Use of drugs that alter the balance;
* Alcohol consumption in the previous 24 hours.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2015-08-10 (Actual); Study Completion 2015-10-03 (Actual)

PRIMARY OUTCOMES:
Evaluation of the sense of joint position. | Before of the application of the protocol exercises
  The sense of joint position was achieved by means of the isokinetic dynamometer (Biodex System 3) triggered in Proprioception mode. Then, the knee joint of each volunteer was slowly extended by the examiner, next to the equipment, at a speed of 20 ° per second, starting from an angle of 90 ° flexion, to the predetermined extension angles: 60 ° and 30 °. With vision occlusion, each volunteer was instructed to memorize the angle, within ten seconds, and then return to the same angle for three attempts.
Evaluation of the muscular electrical activity (Surface electromyograph) of the muscles long fibular, medial gastrocnemius, vastus medialis and gluteus medius . | Before of the application of the protocol exercises
  For the acquisition of electromyographic data, the 8-channel electromyograph was used. The muscles evaluated were the long fibular, the medial gastrocnemius, the vastus medialis and the gluteus medius. Sinak was added for 20 seconds.
Evaluation of the Postural oscillation | Before of the application of the protocol exercises
  The signal for the ground reaction force was acquired by a force platform, which gave the values related to the Vertical Reaction Force of the volunteers. For this, the vertical force platform EMG System do Brasil, model BIOMEC400 was used.
  During the evaluation, the subjects reproduced the unipodal support position over the non-dominant lower limb with the contralateral limb in a knee flexion near 90 ° within 20 seconds. The equipment was installed on a solid and flat base to avoid undesirable vibrations and displacement during the application of forces on the upper surface.

SECONDARY OUTCOMES:
Evaluation of the sense of joint position | After one exercise session (after 1º day of treatment)
  The sense of joint position was achieved by means of the isokinetic dynamometer (Biodex System 3) triggered in Proprioception mode. Then, the knee joint of each volunteer was slowly extended by the examiner, next to the equipment, at a speed of 20 ° per second, starting from an angle of 90 ° flexion, to the predetermined extension angles: 60 ° and 30 °. With vision occlusion, each volunteer was instructed to memorize the angle, within ten seconds, and then return to the same angle for three attempts.
Evaluation of the muscular electrical activity of the muscles of the long fibular, the medial gastrocnemius, the vastus medialis and the gluteus medius | After one exercise session (after 1º day of treatment)
  For the acquisition of electromyographic data, the 8-channel electromyograph was used. The muscles evaluated were the long fibular, the medial gastrocnemius, the vastus medialis and the gluteus medius. Sinak was added for 20 seconds.
Evaluation of the Postural oscillation | After one exercise session (after 1º day of treatment)
  The signal for the ground reaction force was acquired by a force platform, which gave the values related to the Vertical Reaction Force of the volunteers. For this, the vertical force platform EMG System do Brasil, model BIOMEC400 was used.
  During the evaluation, the subjects reproduced the unipodal support position over the non-dominant lower limb with the contralateral limb in a knee flexion near 90 ° within 20 seconds. The equipment was installed on a solid and flat base to avoid undesirable vibrations and displacement during the application of forces on the upper surface.

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda PS Lima, Researcher, Study Director — Universidade do Vale do Paraíba
Locations (1):
- Laboratório de Engenharia de Reabilitação Sensorio Motora, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No